CLINICAL TRIAL: NCT01111734
Title: N-Acetylcysteine in the Treatment of Deliberate Self-Harm in Adolescents: An Open Label Pilot Study
Brief Title: Early Study of N-Acetylcysteine to Treat Deliberate Self-Harm in Adolescents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Minnesota Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0909M72855
Record Dates: First submitted 2010-04-26; First posted 2010-04-28 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Deliberate Self Harm
Keywords: self harm; self injury; self mutilation; N-Acetylcysteine; adolescents; impulse control disorder; borderline personality disorder; fMRI
MeSH Terms: conditions — Self-Injurious Behavior; Self Mutilation; Disruptive, Impulse Control, and Conduct Disorders; Borderline Personality Disorder | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Group (Experimental): The study consists of eight weeks of open label N-Acetylcysteine. All eligible study subjects will be treated with 600mg of N-Acetylcysteine twice a day for 2 weeks, then the dose will be increased to 1200mg twice a day for two weeks, and to 1800mg twice a day for 4 weeks. weeks. Subjects will be seen every two weeks during the 8-week study. Efficacy and safety assessments will be performed at each visit.
  Interventions: Dietary Supplement: N-Acetylcysteine; Drug: fMRI
- Control (Experimental): 40 healthy age-matched peers with undergo the same baseline testing as the NAC subjects as well as baseline fMRI. They will not engage in any follow up visits.
  Interventions: Drug: fMRI

INTERVENTIONS:
Dietary Supplement: N-Acetylcysteine — All eligible study subjects will be treated with 600mg of N-Acetylcysteine orally twice a day for 2 weeks, then the dose will be increased to 1200mg twice a day for two weeks, and to 1800mg twice a day for 4 weeks.
  Other Names: NAC, N-Acetylcysteine; Brand: Swansons Vitamins; 600mg capsule
  Arms: Treatment Group
Drug: fMRI — All eligible subjects and controls will undergo an emotional face-viewing task in our fMRI paradigm in order to focus in on the circuitry related to affect processing.
  Other Names: Seimens 3T MRI

SUMMARY:
Deliberate Self-Harm (DSH) among adolescents is a serious behavioral problem associated with significant injury, impaired functioning, reduced quality of life, and high rates of psychiatric hospitalizations. While DSH has not been shown to have a direct link to suicide attempts themselves, there is a clear link between individuals who engage in DSH and overall rates of suicide. There is currently no medication treatment approved by the FDA for the treatment of DSH.

The goal of this study is to evaluate the efficacy and safety of the dietary supplement N-Acetylcysteine in adolescents aged 13-21 with deliberate self-harm behaviors. There will be an additional neuroimaging component to expand knowledge regarding the neural correlates of this treatment in the study population. We hypothesize that N-Acetylcysteine will reduce the severity of deliberate self harm behaviors because this supplement has been helpful in treating disorders that share some similar traits with DSH. We will be using this medication in 40 young people who deliberately harm themselves and we will assess the severity of their behaviors while being treated with this dietary supplement. We also will collect neuroimaging data on the study participants at baseline and after the treatment with N-Acetylcysteine and compare it to 40 age-matched healthy peer neuroimaging data. The purpose of including this healthy group is to expand knowledge about neural correlates of the study population prior to treatment.

DETAILED DESCRIPTION:
Deliberate Self-Harm (DSH) among adolescents is a serious behavioral problem associated with significant morbidity and mortality, impaired functioning, reduced quality of life, and high rates of psychiatric hospitalizations. Rates of DSH among high-school adolescents range between 14% and 21%, highlighting the need for effective behavioral and pharmacological interventions . Because DSH has been closely linked to Borderline Personality Disorder (BPD), treatments that have been used successfully for BPD such as Dialectical Behavior Therapy (DBT) have been used to treat adolescents with DSH. While DSH has not been shown to have a direct link to suicide attempts themselves, there is a clear link between individuals who engage in DSH and overall rates of suicide. In addition to these high rates of DSH in adolescents, research is continuing to show that similar to adult patients; adolescent DSH is related to high levels of impulsivity.

Considerable advances in the understanding of the neurobiology of risk and reward and impulsivity have improved the general understanding of the neuropathology of a behavior such as DSH. Our previous neuroimaging research of DSH in BPD found that frontal white matter integrity was significantly impaired in these individuals. One conceptualization of DSH is that it represents an imbalance between a strong desire for the reward of DSH (i.e. an overactive ventral tegmental area [VTA]) and an inability to inhibit the drive (i.e. impaired inferior frontal cortex). If the frontal cortex is impaired due to inadequate white matter integrity as our earlier study demonstrated, then reducing the drive for DSH may be the most beneficial target for treatment. Glutamate is known to activate dopamine neurons in the VTA. Because such activation can increase dopamine release in mesocorticolimbic targets, this glutamate-dopamine interaction in the VTA may underlie the chronic reward-seeking that underlies DSH. In fact, dysregulated prefrontal cortex-nucleus accumbens synaptic glutamate transmission appears to underlie the unmanageable motivation to engage in DSH.

Because interactions of glutamate with the dopaminergic system within the VTA mediate reward, N-acetyl cysteine (NAC), a glutamate modulating agent, should attenuate the rewarding properties of DSH by interfering with DSH-induced stimulation of the mesolimbic dopaminergic pathway. NAC increases the activity of cysteine-glutamate antiporters in the nucleus accumbens and abolishes reward-seeking behavior. Behaviorally, NAC administration should lead to diminished urges to engage in DSH. Increased extracellular glutamate by NAC may correct the underlying pathophysiology and symptoms of this compulsive drive to self-injure. NAC has been extensively studied in a variety of medical problems (e.g., cocaine dependence, acetaminophen overdose, AIDS, gambling), and its lack of significant side effects may present a marked advantage over pharmacological agents.

There is a need to develop effective treatment options that are well tolerated, widely available, and do not have prohibitive costs. NAC is an amino acid, available in health food stores, cheaper than the cost of most insurance co-payments, and is easily tolerated. If effective, NAC could be a treatment option available to people throughout the country that do not currently have insurance but are suffering from DSH.

The population to be studied for this trial is 40 men and women, ages 13-21, who engage in deliberate self-harm behaviors at least twice a month. We will also add a sample of 40 matched healthy adolescents to serve as a comparison group for the baseline neuroimaging measures. Study participants will be recruited from outpatient mental health clinics and from the community through advertisements.

The study consists of two components: treatment with N-acetyl cysteine and brain imaging. Participants will be invited to participate in either or both, depending on the distinct eligibility criteria of the two components (see below.)

Treatment component:

The treatment component of the study consists of eight weeks of open label N-Acetylcysteine (NAC). All eligible study subjects will be treated with 600mg of NAC twice a day for 2 weeks, then the dose will be increased to 1200mg twice a day for two weeks, and to 1800mg twice a day for 4 weeks. weeks. Subjects will be seen every two weeks during the 8-week study. Efficacy and safety assessments will be performed at each visit.

Imaging component: A brain imaging session will take place before and after the treatment with NAC. For individuals that either chose not to compete the treatment component or who did not meet entry criteria, they will only have the baseline scan.

The healthy group will only participate in assessment and neuroimaging, not in the treatment or the second scan.

All participants will undergo a comprehensive clinical assessment which will include the following interviews/rating scales/tests:

1. KSADS interview (adolescents and parents) or SCID (adult participants)
2. Child Depression Rating Scale-Revised (CDRS-R)
3. Columbia Suicide Severity Rating Scale (CSSRS) (patients only)
4. Inventory of Statements About Self-Harm (ISAS) (patients only)
5. The Deliberate Self Harm Inventory (DSHI) (patients only)
6. Deliberate Self Harm Questionnaire (DSHQ) (patients only)
7. Beck Depression Inventory-II (BDI-11)
8. Wechsler Abbreviated Scale of Intelligence (WASI)
9. Edinburgh Handedness inventory
10. Iowa Gambling Task (IGT)
11. NIH Toolbox
12. Tanner Questionnaire
13. Eating Questionnaire (EDEQ)
14. Personality Assessment Inventory (PAI)
15. Symptom Check-List-90-R (SCL-90)
16. Barrett Impulsivity Scale (BIS)
17. Difficulties in Emotion Regulation Scale (DERS)
18. Satisfaction with Life Questionnaire
19. Toronto Alexithymia scale
20. Rejection Sensitivity Questionnaire - Adolescent (RSQ-A)

All participants will be invited to undergo an MRI session that includes a structural scan, a resting state fMRI scan, an emotion task fMRI scan, diffusion tensor imaging, and magnetic resonance spectroscopy in the anterior cingulate cortex.

Every two weeks the following assessments will be utilized to assess the efficacy of current treatment on NAC participants:

1. Inventory of Statements About Self-Injury Since Last Visit version (ISAS - SLV)
2. Self-Injury Assessment Scale (SIAS)
3. Deliberate Self Harm Inventory Clinical Change Version (DSHI - CCV)
4. Columbia Suicide Severity Rating Scale Since Last Visit version (CSSRS - SLV)

At the end of the 8 week administration of NAC participants will complete:

1. Inventory of Statements About Self-Injury Since Last Visit version (ISAS - SLV)
2. Self-Injury Assessment Scale (SIAS)
3. Deliberate Self Harm Inventory Clinical Change Version (DSHI - CCV)
4. Columbia Suicide Severity Rating Scale Since Last Visit version (CSSRS - SLV)
5. Barrett Impulsivity Scale (BIS)
6. SCL-90
7. DERS
8. Satisfaction with Life Questionnaire
9. BDI-II
10. Iowa Gambling Task (IGT)
11. The same MRI protocol as described above.

ELIGIBILITY:
Inclusion Criteria:

All participants:

1. Participants must be aged 13 years to 21 years with the ability to provide consent or guardian consent and assent.
2. They must be available to come to the University of Minnesota for study visits.

All DSH participants:

1) Must have engaged in DSH at least 4 times, with most recent episode in past three months.

Controls

1. Have no history of deliberate self-harm
2. Have no current or past psychiatric diagnoses

Exclusion Criteria:

1. Those who are pregnant, breastfeeding, or who have a positive urine drug screen will not be included.
2. Individuals with unstable medical illnesses, a history of seizures or heart attack, or arrhythmia not be included.
3. Participants will not have a history of Bipolar type I or II, dementia, schizophrenia or any other psychotic disorder.
4. Patients with active suicidal intent will not be included.
5. If DSH participants are currently taking medications, the doses of these must be stable 1 month prior to study onset.

For Receiving NAC:

1. Participants may not be taking the following medications concurrently, due to the possibility of medication interactions: activated charcoal, ampicillin, carbamazepine, cephaloridine, cloxacillin, methicillin, nitroglycerin, oxacillin, penicillin G, quinacillin.
2. Participants cannot have a history of allergic reaction to NAC.

For MRI Scanning:

1. Participants may not have any metal in their body that would be unsafe in an MRI scanner.
2. Participants with claustrophobia will not be included.

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 67 (Actual)
Dates: Start 2011-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Deliberate Self Harm Inventory Clinical Change Version (DSHI-CCV) | Every 2 weeks
  Assesses frequency and type of deliberate self harm.
K-SADS-PL | Intake
  A semi-structured clinical interview conducted separately with child and parent. Clinicians formulate the diagnosis during a consensus meeting, combining all clinical information.
Inventory of Statements about Self-Injury (ISAS) | Every 2 weeks
  Questionnaire regarding self injurious behavior.

SECONDARY OUTCOMES:
Columbia Suicide Severity Rating Scale (CSSRS) | Every 2 weeks
  Measure of suicide risk to assess safety during the study.
Barrett Impulsivity Scale (BIS) | Intake, Exit
  This instrument will assess the effect of the intervention on impulsivity factors.
Deliberate Self-Harm Questionnaire-Mood (DSHQ-M) | Intake
  Questionnaire regarding mood before, after, and during engaging in self-injurious behavior.
BDI-II | Intake, Baseline MRI, Exit MRI
  Assesses depressive mood in last two weeks.
Iowa Gambling Task (IGT) | Intake, Exit
  Game used to measure reward processing
Symptom Check-List 90 (SCL-90) | Intake, Exit
  Looks at correlation between amygdala-thalamus connectivity and interpersonal sensitivity.
Difficulties in Emotion Regulation Scale (DERS) | Intake, Exit
  Used to assess capacity for emotion regulation.
Children's Depression Rating Scale - Revised (CDRS-R) | Intake
  A questionnaire that will help assess participant's depression
NIH Toolbox | Intake
  The NIH tool box is compromised of 2 computer-based measures: the Flanker Task, and the Dimensional Card Sort Test. The participant will complete both measures. These will measure neurocognitive functioning
Wechsler Abbreviated Scale of Intelligence (WASI-2) | Intake
  Used to assess IQ
Tanner Questionnaire | Intake
  This questionnaire will be used to assess pubertal stages of participants
Personality Assessment Inventory (PAI) | Intake
  A multi-scale test of psychological functioning that assesses constructs relevant to personality and psychopathology evaluation.
Satisfaction with Life Scale | Intake, Exit
  This questionnaire looks at the participants satisfaction with their life at the moment
Toronto Alexithymia Scale (TAS) | Intake, Exit
  Will assess the presence or extent to which the participant exhibits Alexithymia.
Rejection Sensitivity Questionnaire - Adolescent (RSQ-A) | Intake
  Assesses the extent to which the participant perceives rejection in their daily lives.
Self-Injury Assessment Scale (SIAS) | Every 2 weeks
  Provides more information about the participant's self-harm behaviors over the past two weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn R Cullen, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Dept. of Psychiatry Ambulatory Research Center, Minneapolis, Minnesota, United States